CLINICAL TRIAL: NCT00627562
Title: A Pilot Study of the Use of the DaVinci Robotic System for Otorhinolaryngology-Head and Neck Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Richard V. Smith, MD, Vice Chairman, Otorhinolaryngology/head and neck surgery, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-03-080
Record Dates: First submitted 2008-02-05; First posted 2008-03-03 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Neoplasms
Keywords: robotic; robot assisted; minimally invasive; tumors of head and neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): robot assisted endoscopic head and neck surgery
  Interventions: Device: robot assisted endoscopic head and neck surgery using the DaVinci Robotic Surgical System

INTERVENTIONS:
Device: robot assisted endoscopic head and neck surgery using the DaVinci Robotic Surgical System — Planned endoscopic surgery of the head and neck performed with the DaVinci Robotic Surgical System

SUMMARY:
1. Patients included will have benign or malignant lesions with treatment plan for endoscopic resection or resection by other minimally invasive techniques.
2. They will be offered a robotic approach to their surgery using the DaVinci robotic surgical system (intuitive Surgical, Inc.).
3. The objectives are to evaluate our ability to adequately visualize the surgical field and perform the intended surgery without a higher complication rate.
4. Secondary objective include evaluation of blood loss, length of hospital stay, complications while using the DaVinci robot system, and quality of life in subjects and historical controls undergoing similar surgery without the robot or radiation therapy.
5. To evaluate recurrence, survival and other outcome data in robotic surgery patients compared with similar historical control groups (matched with respect to stage, prior and subsequent treatment, age, tumor HPV positivity) of patients who have undergone standard surgery without the robot or radiation/chemoradiation treatment as an alternative to surgery.

5. Endpoints will be compared to historical controls.

DETAILED DESCRIPTION:
The da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) being evaluated in this pilot study consists of 3 basic components: a surgeon's console, articulated mechanical arms and sterilizable instruments. The console includes a computer, video monitor and instrument controls, and is located in the operating room adjacent to the operating room table. The console is connected via computer to the mechanical arms holding the endoscope (surgical TV camera) and sterile surgical tools (e.g., forceps, scissors, electrocautery, etc.). These arms are located immediately adjacent to the patient on the operating room table. The surgeon sits at the console and controls the position and movement of the arms and surgical tools. The design of these tools is based upon well-established, commonly used surgical instruments. The da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) is a "manual image-guided surgery" system that is computer enhanced rather than "computer guided robotic surgery" in which the surgeon programs the computer to do the surgery and the robot does the surgery (also known as a "milling" device).22 Use of the da Vinci® Robotic Surgical System (Intuitive Surgical, Inc., Sunnyvale, CA) in the aforementioned configuration in fact facilitates an exact translation of the surgeon's hand and finger movements at the console to precise and tremor-free movements of the arms and instruments.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years f age
* Indications for diagnostic or therapeutic approaches for benign or malignant disease of the head and neck
* Written informed consent

Exclusion Criteria:

* Unexplained fever and/or untreated, active infection
* Pregnancy
* Previous head and neck surgery precluding transoral/endoscopic/robotic procedures
* Presence of medical conditions contraindicating general anesthesia or transoral surgical approaches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-07; Primary Completion 2014-06 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
ability to adequately visualize the operative field and complete planned surgery | 1 day

SECONDARY OUTCOMES:
complication rate compared to standard endoscopic and minimally invasive procedures | 1 month
blood loss compared to historical controls of endoscopic and minimally invasive procedures | 1 day
quality of life at early (1-3 months) and late (one year) | 1 year
number of days hospitalized immediately after surgery | at discharge from hospital
Time to recurrence of tumor or other pathology for which procedure was performed | at recurrence of tumor or pathology
Time from start of treatment to death | at time of death

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Smith, MD, Study Chair — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Gourin CG, Terris DJ. Surgical robotics in otolaryngology: expanding the technology envelope. Curr Opin Otolaryngol Head Neck Surg. 2004 Jun;12(3):204-8. doi: 10.1097/01.moo.0000122309.13359.af. PMID 15167030
- [Background] Hockstein NG, Nolan JP, O'Malley BW Jr, Woo YJ. Robot-assisted pharyngeal and laryngeal microsurgery: results of robotic cadaver dissections. Laryngoscope. 2005 Jun;115(6):1003-8. doi: 10.1212/01.WNL.0000164714.90354.7D. PMID 15933510
- [Background] Hockstein NG, O'Malley BW Jr, Weinstein GS. Assessment of intraoperative safety in transoral robotic surgery. Laryngoscope. 2006 Feb;116(2):165-8. doi: 10.1097/01.mlg.0000199899.00479.75. PMID 16467698
- [Background] Lobe TE, Wright SK, Irish MS. Novel uses of surgical robotics in head and neck surgery. J Laparoendosc Adv Surg Tech A. 2005 Dec;15(6):647-52. doi: 10.1089/lap.2005.15.647. PMID 16366877
- [Background] Tanna N, Joshi AS, Glade RS, Zalkind D, Sadeghi N. Da Vinci robot-assisted endocrine surgery: novel applications in otolaryngology. Otolaryngol Head Neck Surg. 2006 Oct;135(4):633-5. doi: 10.1016/j.otohns.2006.07.003. No abstract available. PMID 17011430